CLINICAL TRIAL: NCT04301895
Title: Pupillary Unrest in Ambient Light, and Relationship to Opioid-Induced Respiratory Depression in Volunteers
Brief Title: Pupillary Unrest in Ambient Light, and Relationship to Opioid-Induced Respiratory Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 221163
Record Dates: First submitted 2020-03-03; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Opioid; Intoxication, Perception Disturbance (Acute); Acute Pain; Overdose of Opiate; Respiratory Depression; Safety Issues
MeSH Terms: conditions — Acute Pain; Opiate Overdose; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Each subject is his/her own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interactive (Other): Subject will be asked to continually interactive with the investigators, answering a series of standard questions during the remifentanil infusion and recovery periods.
  Interventions: Behavioral: Continuous conversational interaction; Drug: Remifentanil infusion
- Non-interactive (Other): All verbal interaction will be avoided and extraneous sounds will be eliminated from the environment during the remifentanil infusion and recovery periods.
  Interventions: Drug: Remifentanil infusion

INTERVENTIONS:
Behavioral: Continuous conversational interaction — Maintaining continuous conversation, requiring that the subject answer questions and engage in discussion without interruption.
  Other Names: Environmental stimulation
  Arms: Interactive
Drug: Remifentanil infusion — 10 minute remifentanil infusion

SUMMARY:
Volunteers will receive a weight-based opioid (remifentanil) infusion for 10 minutes. In the first run, serial pupillary measurements (pupillary unrest, pupil diameter) will be taken at baseline, and at 2.5-minute intervals during the infusion and a 25-minute recovery period afterwards. After a washout period, the experiment will be repeated in each subject (second run). The two runs differ only by presence versus absence of verbal interaction.

DETAILED DESCRIPTION:
Healthy volunteers aged 20-55 will receive a weight-based opioid (remifentanil) infusion for 10 minutes. Vital signs including SpO2, transcutaneous CO2, and respiratory rate will be continuously measured.

In the first run, serial pupillary measurements (pupillary unrest, pupil diameter) will be taken at baseline, and at 2.5-minute intervals during the infusion and a 25-minute recovery period afterwards. After a washout period, the experiment will be repeated in each subject (second run). The two runs differ only by presence of ongoing verbal interaction versus complete avoidance of verbal interaction.

Incidence of respiratory depression will be compared in the two protocols with or without verbal interaction. Correlation between pupil diameter and pupillary unrest with estimated opioid concentrations will be determined by regression. Difference between pupil measurement versus opioid concentration regressions will be compared by chi2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Able to provide informed consent

Exclusion Criteria:

* Active substance use disorder
* Prior opioid use disorder
* Opioid use within 30 days.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Impact of environmental stimulation on decline in oxygen saturation to ≤ 90%. | 35 minutes
  Conversational interaction and oxygen saturation measured by pulse oximeter.
Impact of environmental stimulation on CO2 increase of 15% or more above baseline. | 35 minutes
  Conversational interaction and CO2 measured by transcutaneous sensor.
Correlation between estimated opioid concentration and deviation in pupillary measurement. | 35 minutes
  Relationship of opioid concentration to pupillary unrest, measured by the pupillometer

SECONDARY OUTCOMES:
Impact of environmental stimulation on opioid-related deviations in pupillary measurements. | 35 minutes
  Impact of conversational interaction on degree of decline in pupillary unrest as measured by the pupillometer.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Eshima McKay, M.D., Principal Investigator — Professor of Anesthesia
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKay RE, Kohn MA, Larson MD. Pupillary unrest, opioid intensity, and the impact of environmental stimulation on respiratory depression. J Clin Monit Comput. 2022 Apr;36(2):473-482. doi: 10.1007/s10877-021-00675-3. Epub 2021 Mar 2. PMID 33651243